CLINICAL TRIAL: NCT00515944
Title: Evaluate the Migration Potential of Xeomin® Compared to Two Other Botulinum Toxin Type A Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Clinical Pharmacology, Merz Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: MRZ 60201-0709/1
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: No condition; healthy volunteers
MeSH Terms: interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum neurotoxin type A, free of complexing proteins

SUMMARY:
Xeomin® is a Botulinum neurotoxin type A preparation free of complexing proteins, i.e. free of bacterial proteins other than the active toxin. Injected into the muscle, Xeomin® causes local weakening. Botulinum toxin type A is used for certain neurological and aesthetic treatments. This study will investigate the migration potential of Xeomin®.

DETAILED DESCRIPTION:
Conducted in Europe

ELIGIBILITY:
Inclusion Criteria:

* Healthy females, 18 to 65 years

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Measurement of area

CONTACTS AND LOCATIONS:
Overall Officials: Merz Pharmaceuticals, Study Chair — Merz Pharmaceuticals GmbH
Locations (1):
- Merz Pharmaceuticals GmbH, Frankfurt am Main, Germany